CLINICAL TRIAL: NCT01356095
Title: A Knowledge Translation Intervention for TB/HIV Treatment Adherence, in Zomba District, Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dignitas International (Other)
Collaborators: University of Toronto (Other); Ministry of Health and Population, Malawi (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DI807
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2011-05

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Treatment Adherence; knowledge translation; Educational outreach
MeSH Terms: conditions — Tuberculosis; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PALM-Plus control (Active Comparator): Health centers randomized to Palm-Plus intervention in larger trial this trial is embedded in, but not receiving the adherence intervention.
  Interventions: Other: Palm-Plus
- Adherence intervention (Experimental): Intervention arm.
  Interventions: Other: Knowledge translation intervention
- Control (No Intervention)

INTERVENTIONS:
Other: Knowledge translation intervention — Two part intervention includes an educational outreach intervention for health care workers and a point of care patient education/counselling tool, delivered to providers within health centers randomized to the intervention arm, using a train the trainer on-site training model.
  Arms: Adherence intervention
Other: Palm-Plus — Clinical guideline and training approach, designed for mid-level healthworkers.
  Arms: PALM-Plus control

SUMMARY:
Despite increased emphasis on evidence based practice in recent years a gap remains between evidence and practice, particularly in resource poor countries. Few studies to date have examined the use of knowledge translation strategies to improve health care outcomes in low income countries. However, given that the majority of health care in these settings is provided by workers with less training and limited resources, the theoretical potential for knowledge translation strategies to improve health care delivery and outcomes by integrating best evidence into routine practice may be greatest in these settings.

Knowledge translation (KT) is an approach to changing health care provider behavior to reduce the gap between evidence and practice in health care delivery. There has been a tendency for knowledge translation interventions to employ generic, "off the shelf", strategies, and apply them to deal with specific issues. This generic approach, fails to recognize the variability in the specific characteristics of health care settings, in terms of their patient populations, health care systems, and health care providers. These characteristics, whether they function as barriers or facilitators to change, make a generalized approach to KT ineffective, where a tailored strategy, which specifically adjusts its approach to measured local barriers and facilitators may achieve better alignment of practice to evidence. This is likely to be particularly true in low income countries where the majority of health care is provided by non-physician health care workers, working within a wider range of health care systems, with variable and unique patient populations and resource constraints. Given the potential to significantly impact health care outcomes at relatively low cost, further research is needed both to develop methods for identifying potential barriers and facilitators to KT strategies in specific resource poor settings, and to evaluate the effectiveness of KT strategies tailored to address the identified barriers.

This study will assess the effectiveness of a two part knowledge translation intervention tailored to address factors identified in a previous study as functioning as barriers and facilitators to treatment adherence among patients on treatment for tuberculosis or combined tuberculosis and antiretroviral treatment, targeting improved patient adherence and health outcomes, in a specific low income country.

ELIGIBILITY:
Inclusion Criteria:

* All health centers in Zomba District

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients classified as successfully treated. | 1 year
  Treatment success is defined as cure or treatment completion. Outcomes measured at patient level at end of treatment (6 months), and at 1 year at health center level (randomized at level of health center)

SECONDARY OUTCOMES:
Proportion of patients defaulting from treatment. | 1 year
  Default defined as missing greater than or equal 2 consecutive months of treatment. Outcome measured at patient level at end of treatment (6 months), and 1 year at level of health center (randomized at level of health center).
Proportion of successfully treated and default cases among patients treated for tuberculosis only and those on both tuberculosis and antiretroviral treatment | 1 year
  Treatment success defined as cure or treatment completion. Outcome measured at patient level at end of treatment (6 months), and at 1 year for the the health center (randomized at level of health center)
Weight change. | 1 year
  Weight change from start to end of treatment. Outcome measured at patient level throughout treatment (6 months) and at 1 year at the health center level (randomized at level of health center).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Puchalski Ritchie, Principal Investigator — University of Toronto
Locations (1):
- Zomba District Health Centers, Dignitas International, Zomba, Malawi

REFERENCES:
- [Derived] Puchalski Ritchie LM, Schull MJ, Martiniuk AL, Barnsley J, Arenovich T, van Lettow M, Chan AK, Mills EJ, Makwakwa A, Zwarenstein M. A knowledge translation intervention to improve tuberculosis care and outcomes in Malawi: a pragmatic cluster randomized controlled trial. Implement Sci. 2015 Mar 28;10:38. doi: 10.1186/s13012-015-0228-y. PMID 25890186